CLINICAL TRIAL: NCT04092023
Title: Effects of a Self-care Management Programme for Type 2 Adult Diabetic Patients With Poor Glycemic Control in General Out-patients Clinics - a Randomized Control Trial
Brief Title: Self-care Management Programme for Type 2 Adult DM Patients With Poor Glycemic Control
Acronym: T2DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chan Ching Yee, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ChanCY_RP1
Record Dates: First submitted 2019-09-12; First posted 2019-09-17 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nursing Education Research

STUDY DESIGN:
Intervention Model Description: A six month and two-arm parallel randomized control trial is employed
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Participants in control group will be received usual care. They will be gone through yearly DM complication screening. A screening report and information sheet on general DM management will be issued to participants. Therapeutic goals will be set and further conventional health care education intervention will be referred.
  Interventions: Other: nursing education
- Intervention group (Other): The interventions are designed to address the seven key self-management behaviours identified by the Association of American Diabetes Educations: (1) healthy eating, (2) being active, (3) monitoring, (4) taking medication, (5) problem solving, (6) reducing risk, and (7) healthy coping. In addition, the Chronic Care Model elements of self-management support and patient centered-care approach is embraced during the intervention process. The nursing care components provided to participants will be included (a) self-care management knowledge, (b) skill-based learning and problem solving, (c) participants' participation and engagement, (d) participants' in goal setting, and (e) coordinate care, involve participants to make decision.
  Interventions: Other: nursing education

INTERVENTIONS:
Other: nursing education — Participants will be recruited to attend 2 group sessions; each group will have 10-12 participants and each session will be lasted for 120 minutes. Two subsequent phones follow up to participants will be arranged.

SUMMARY:
Type 2 diabetes becomes the most prevalence chronic disease worldwide. Most type 2 diabetes patient are under the care in public general out-patient clinic in Hong Kong. The chronic nature of diabetic and the complexity of its management, on top of medication, diabetic patients often require behaviour modification and self-care management support. Effective diabetes self-care management education with patient-centered care approach with patients' participation and engagement has been shown to improve the clinical outcome. But such application during doctors' consultation are minimal in view of time limitation. Primary Care Nurse (PCN) is the first contact and is easily accessible in GOPCs. With support and training, PCN could act as a case manager to deliver the coordinated care. Interact and engage type 2 diabetes patients in self-care management, and work with multidisciplinary team in providing patient-centered care in GOPC setting. As there is lack of evidence about adopting such approach in the investigator's local population. This study is to test the effectiveness of the PCN led self-care management program to improve patients' clinical outcomes.

DETAILED DESCRIPTION:
1. Safety Assessment

   There is no harmful effect from the intervention.
2. Statistics

   (A) Sample Size Estimation With reference from previous study (Aanand et al. 2011), the sample size is calculated by assuming change the reduction of HbA1c is 0.59% (intervention group 8.05% (SD 1.40) versus control group 8.64% (SD 1.39). In order to have 80% power and 5% false positive error, a sample size of 88 is needed for each arm using the public domain sample size calculator (https://www2.ccrb.cuhk.edu.hk/stat/). After consideration of 10% attrition rate, 97 participants will be recruited in each arm.

   (B) Data Analysis All statistical analyses will be performed using SPSS Windows 22.0 program. P-value less than 0.05 will be considered statistically significant. All treatment evaluations will be performed on the principle of intention-to-treat analysis of the difference in outcomes between groups at 6 months after baseline. Missing values will be imputed using last value carrying forward method. Repeated analysis will be done for per-protocol analysis. Demographics and baseline characteristics will be summarized using descriptive statistics. Continuous variable will be summarized as numbers of observed values, mean and standard deviation. Categorical variables will be described as frequency and percentage. Information collected on all outcomes will be first summarized using descriptive statistics at baseline and at 6 months as appropriate. Linear regression model will be used to test the effect of intervention on the outcomes between 2 groups.
3. Direct Access to Source Data and Documents

   Apart from the outpatient number and Initials, no subject sensitive identifier will be contained in the completed questionnaires. All completed questionnaires will be kept in knocked administrative room in research site with limited access by investigators. All patient records in CMS will be accessed by investigators only by their own CMS login.
4. Quality Control and Quality Assurance

   Expert panel including family medicine specialist, diabetes nurse consultant, diabetes nurse working in primary health care setting, dietitian, physiotherapist and podiatry will review the education contents. Nurses who have received structural education on chronic disease management as organized by Institute of Advanced Nursing Studies, Hospital Authority will be assigned to provide intervention to participants. All the interventionist and co-investigator will be trained for 4 hours by principal investigator for the objectives, contents and process of program before implementation. Meeting will be held during the process of data collection to exchange ideas and knowledge between the interventionist.

   Principal investigator will monitor in all study phase. The interaction between interventionists and participants will be guided by protocol and guideline. Co-investigator in individual clinic will monitor participants' recruitment and data collection. Principal investigator will randomly check and sit in to monitor the consistency.
5. Ethics and Data Handling

Ethics of this study will be complied with the Declaration of Helsinki. Investigators will explain the study in detail and subjects will sign an informed consent form with written information sheet. Investigators will clarify all the queries with subjects. The enrolment will be entirely voluntary and it will not affect their care received in the study site. All the personal identifiers will be removed during data processing. The relevant documents will be kept in a locked cabinet in the study site and will be retained for 3 years after the study end.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >=18
2. Clinically diagnosed of type 2 diabetes
3. Poorly glycemic control with recent HbA1c ≧ 7.5%
4. Chinese participants who could speak Cantonese

Exclusion Criteria:

1. Unable to perform self-care management due to physical or mental limitation
2. Engage in another similar program
3. Pregnancy
4. Life expectancy <1 year due to malignancies or other terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Glycemic control | Assess change from Baseline HbA1c at 6 months
  Blood test for HbA1c

SECONDARY OUTCOMES:
Diabetes Knowledge | Assess change from Baseline HbA1c at 6 months
  The Diabetes Knowledge Scale (DKN) (Dunn et al, 1984) will be adopted to measure participants' knowledge level. The DKN questionnaire consists 15 multiple-choice items each related to test the participants' knowledge level on the major areas of basic physiology of diabetes and general principles of diabetes care. A score of 1 is assigned for a correct response and 0 for an incorrect response. The total score is calculated by summing the scores from 15 items. The total scores are then converted to percentages. High scores on this measure indicated a higher level of diabetes knowledge. The original English version of the DKN questionnaire was translated into Chinese version by Chan & Molassiots (1999) and has been validated for Hong Kong Chinese T2DM patient in an out-patient diabetes clinic. The content validity index is 0.96.
Self-Efficacy: Diabetes Empowerment Scale - Short Form (C-DES-SF) | Assess change from Baseline HbA1c at 6 months
  Diabetes Empowerment Scale - Short Form (C-DES-SF) will be adopted to measure participants' self-efficacy level. It has been validated for Hong Kong Chinese patient by Shiu, Choi & Wong (2012). The Internal consistency (α = 0.77) and the test-retest validity (ICC 0.89, 95% CI 0.86-0.92). The scale consists of 10 items and reports in a 5-points Likert scale. An item checked "strongly agree" receives 5 points; "agree" - 4 points; "neutral" - 3 points; "disagree" - 2 points; and "strongly disagree" receives 1 points. An overall score for the C-DES-SF would be calculated by adding all of the item points. Higher points represent higher level of self-efficacy to manage diabetes in his/her daily live.The items to be reported are (a) overcoming barriers, (b) determining suitable methods, (c) achieving goals, (e) obtaining support, and (f) coping.
QOL: Audit of Diabetes Dependent Quality of Life (ADDQoL-19) | Assess change from Baseline HbA1c at 6 months
  Audit of Diabetes Dependent Quality of Life (ADDQoL-19) will be used to measure participants' QOL. The Internal consistency (α = 0.81) and the construct validity was proven (Fung & Wong, 2016). The scale consists of 19 diabetes-specific domain items and reports in a 7-points scale. Respondents rate the impact of diabetes on applicable domains on a scale from -3 (maxmium negative impact) to +1 (maximum postive impact). Respondents then rate the importance of those domains for their QOL on a scale from 3 (very important) to 0 (not at all important). Impact ratings are multiplied by the corresponding importance rating to provide a weighted-impact score for each domain from -9 (maximum ngeative impact) to +3 (maximum postive impact). Weighted impact score are summed and divided by the number of applicable domains, to give a overall Average Weighted Impact (AWI) score. Higher AWI scores represent a worse of quality of life as impacted by diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: Ching Y Chan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- KWC FM & PHC, Hospital Authority, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will become availiable in 1Q 2021 and starting 6 months after publication
Access Criteria: Principle investigator will review requests